CLINICAL TRIAL: NCT05152732
Title: Safety and Tolerability of VGB-R04 in Patients With Haemophilia B
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021043
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia B
Keywords: Hemophilia; AAV; safety; gene therapy
MeSH Terms: conditions — Hemophilia B; Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGB-R04 (Experimental): Single intravenous (i.v.) infusion of VGB-R04 Intervention: Gene Therapy / Gene Transfer
  Interventions: Genetic: VGB-R04

INTERVENTIONS:
Genetic: VGB-R04 — A novel, bioengineered adeno-associated viral (AAV) vector carrying human factor IX variant

SUMMARY:
An Open-Label, Non-Randomized, uncontrolled, single-dose pilot study of VGB-R04 in subjects with Hemophilia B.

DETAILED DESCRIPTION:
Hemophilia B is a genetic bleeding disorder caused by pathogenic variants (eg, mutations, deletion) in the FIX gene. HB patients have frequent and potentially life-threatening bleeding and often develop progressive physical disability and pain from chronic haemarthropathy. Current replacement therapy needs regular treatment in the life-long time, bringing heavy economic and social burdens.

VGB-R04 is a novel AAV vector carrying a high specific activity factor IX variant. This study is intended to evaluate the safety, tolerability and kinetics of a single IV infusion of VGB-R04. All subjects in this study will provide informed consent and then undergo screening assessments up to 6 weeks before administration of VGB-R04. All subjects will undergo 52(±2) weeks of safety observation and will be encouraged to enroll in an extension study to evaluate the long-term safety of VGB-R04 for a total of five years.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years and ≤75years of age;
2. Confirmed diagnosis of hemophilia B (baseline FIX activity ≤ 2% of normal or documented history of FIX activity ≤2%);
3. At least 100 days exposure history to FIX;
4. Currently receiving FIX Prophylaxis therapy or on-demand treatment to prevent bleeding;
5. Have acceptable laboratory values:

   1. Hemoglobin ≥110 g/L;
   2. Platelets ≥100×10'9 cells/L;
   3. AST, ALT, alkaline phosphatase ≤2×upper limit of normal (ULN) at the testing laboratory;
   4. Bilirubin ≤3× ULN ;
   5. Creatinine ≤1.5× ULN.
6. No measurable factor IX inhibitor as assessed by the central laboratory and have no prior history of inhibitors to factor IX protein;
7. Agree to use reliable barrier contraception until 3 consecutive samples are negative for vector sequences;
8. Able to provide informed consent and comply with the requirements of the study.

Exclusion Criteria:

1. Have significant underlying liver disease within the past 6 months prior to or at Screening, including but not limited to:

   1. Preexisting diagnosis of portal hypertension;
   2. Splenomegaly;
   3. Encephalopathy;
   4. Reduction of serum albumin;
   5. Evidence of significant liver fibrosis;
2. Have anti-VGB-R04 neutralizing antibody titers ≥1:5;
3. Evidence of severe infection disease, i.e., human immunodeficiency virus (HIV) infection, syphilis, tuberculosis, etc.;
4. Evidence of active hepatitis B virus infection (HBV-DNA >103 IU/ml) or hepatitis C virus infection (HCV antigen and HCV-RNA positive);
5. Evidence of malignant tumours or those with a previous history of malignant tumours;
6. Have a history of chronic infection or other chronic diseases that the Investigator considers to constitute an unacceptable risk;
7. Any immunodeficiency;
8. Participated in a gene transfer trial within the last 52 weeks or in a clinical trial with an investigational drug within the last 4 weeks;
9. Have used glucocorticoids, immunosuppressive drugs, or antipsychotics within the last 3 months;
10. Previous history of hypersensitivity or allergic reaction to any FIX products or any immunoglobulin;
11. Unable or unwilling to comply with the schedule of visits and study assessments described in the clinical protocol;
12. Any concurrent clinically significant major disease or any other condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Baseline up to Week 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of serious adverse events | Baseline up to Week 52
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that resulted in death; life threatening; require inpatient hospitalization or prolongation of existing hospitalization; result in persistent or significant disability/incapacity; result in congenital anomaly/birth defect
Number of Participants with Clinically Significant Change from Baseline in Vital Signs | Baseline up to Week 52
  Vital signs (temperature, respiratory rate, pulse rate, systolic and diastolic blood pressure) will be obtained with participants in the seated position, after having sat calmly for at least 5 minutes. The clinical significance of vital signs will be determined at the investigator's discretion
Number of Participants with Clinically Significant Change From Baseline in Physical Examination Findings | Baseline up to Week 52
  The physical examination will include examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination will assess the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant-reported symptoms. Findings will be considered to be clinically significant based on the investigator's decision
Number of Participants with Clinical Laboratory Abnormalities | Baseline up to Week 52
  Physical examination included examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant-reported symptoms. Findings were considered to be clinically significant based on the investigator's decision.

SECONDARY OUTCOMES:
Vector- derived FIX:C Activity | Baseline up to Week 52
  All samples collected from participants for plasma FIX activity levels will be analyzed and used to determine peak and steady-state vector-derived circulating FIX activity levels
Vector- derived FIX antigen levels | Baseline up to Week 52
  The vector-derived endogenous (not affected by intercurrent FIX product infusions) FIX:C activity antigen levels will be characterized by post-treatment population mean
Annualized bleeding rate changes from baseline | Baseline up to Week 52
  The number of bleeding episodes per participant will be recorded, and the annualized number of bleeding episodes was calculated
Annualized FIX consumption changes from baseline | Baseline up to Week 52
  The use of on-demand FIX replacement therapy will be recorded by dose (IU/kg) administered, and the annualized use of FIX replacement therapy will be calculated.
Number of target joints | Baseline up to Week 52
  The criterion of the target joint is a minimum of three bleeds into a single joint within a consecutive three-month period.
Vector shedding of VGB-R04 | Baseline up to Week 52
  Saliva, urine and semen will be collected to assess clearance of vector genomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Blood diseases hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGB-R04 is fully approved.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be shared with other researchers when VGB-R04 is fully approved.
Access Criteria: IPD will be shared with other researchers when VGB-R04 is fully approved.